CLINICAL TRIAL: NCT00379574
Title: A Phase I/II Study of Bortezomib Plus CHOP Every 2 Weeks in Patients With Advanced Stage Diffuse Large B-cell Lymphomas
Brief Title: Bortezomib Plus CHOP Every 2 Weeks for Advanced Stage DLBCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Principal Investigator, Cheolwon Suh, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2006-276
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Lymphoma, Large-Cell, Diffuse; Lymphoma, B-Cell
Keywords: diffuse large B-cell lymphoma; Bortezomib; CHOP; Lenograstim
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell | interventions — Bortezomib; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; Lenograstim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib + CHOP every 2 weeks (Experimental): Bortezomib + CHOP(Cycloophosphamide, vincristine, doxorubicin,and predinisolone) every 2 weeks
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: Lenograstim

INTERVENTIONS:
Drug: Bortezomib — Bortezomib:
  For phase I, 3 dose levels (1.0, 1.3 or 1.6 mg/m2), days 1 and 4, every 2 weeks.
  For phase II, suggested dose of Bortezomib through phase I, days 1 and 4, every 2 weeks.
  Other Names: velcade
Drug: Cyclophosphamide — cyclophosphamide 750mg/m2 day 1, every 2 weeks
  Other Names: cytoxan
Drug: Doxorubicin — doxorubicin 50 mg/m2 day 1, every 2 weeks
  Other Names: adriamycin
Drug: Vincristine — vincristine 1.4 mg/m2 (max. 2 mg) day 1, every 2 weeks
  Other Names: Oncovin
Drug: Prednisolone — prednisolone 100 mg days 1-5, every 2 weeks
  Other Names: Pd
Drug: Lenograstim — Lenograstim 5 microgram/kg subcutaneously days 4-13 every 2 weeks
  Other Names: Neutrogin; G-CSF

SUMMARY:
Diffuse large B-cell lymphoma is a most prevalent non-Hodgkin's lymphoma. Recently the clinical results have been improved with new drugs and new modalities such as cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) every 2 weeks. Bortezomib is well known to be effective for multiple myeloma and has been being tried for other malignancies including lymphoma. The investigators will incorporate Bortezomib to CHOP every 2 weeks to further improve the clinical efficacy in diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Intended number of patients: 63 patients in total

* Phase I: 9 patients for 3 levels
* Phase II: 50 patients plus 3 patient from Phase I at MTD level
* Plus 4 patients: considering 5% follow-up loss rate

Study design and methodology:

For phase I, 9 patients; 3 levels of bortezomib (1.0, 1.3 and 1.6 mg/m2), 3 patients at each dose level.

If escalation of bortezomib beyond 1.0 mg/m2 is not possible, the trial will be stopped.

For phase II, 53 patients (3 from phase I at MTD level); Reject when complete response rate equal or less than 12/19 or 37/53 by Simon two-stage optimal phase II design.

Treatments:

* Bortezomib:

For phase I, 3 dose levels (1.0, 1.3 or 1.6 mg/m2), days 1 and 4, every 2 weeks.

For phase II, suggested dose of Bortezomib through phase I, days 1 and 4, every 2 weeks.

* CHOP2: cyclophosphamide 750mg/ m2 day 1, vincristine 1.4 mg/ m2 (max. 2 mg) day 1, doxorubicin 50 mg/ m2 day 1, prednisolone 100 mg days 1-5, every 2 weeks.
* G-CSF: Lenograstim 5 microgram/kg subcutaneously days 4-13 every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLBCL
* Age 70 years or less
* Previously untreated
* Performance status: ECOG 0-2
* Advanced stage: stage III, IV, or non-contiguous stage II
* Measurable disease: 1 cm or more by spiral CT
* Normal liver function

Exclusion Criteria:

* Platelet count less than 75,000/microL within 14 days before enrollment.
* Absolute neutrophil count of less than 1,500/microlL within 14 days before enrollment.
* Cr more than 2.0 mg/dL and/or calculated or measured creatinine clearance less than 50 mL/min within 14 days before enrollment.
* Peripheral neuropathy of Grade 2 or worse within 14 days before enrollment.
* Hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding.
* Other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Uncontrolled or severe cardiovascular disease, including MI within 6 months of enrolment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheolwon Suh, M.D.,Ph.D., Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Asan Medical Cener, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Duration of patient enrollment: From 15-Dec-2006 to 02-May-2009
Groups:
- Bortezomib + CHOP Every 2 Weeks: 1. Phase I Bortezomib 1.0, 1/3, and 1.6 mg/m2 CHOP,every 2 weeks cyclophosphamide 750 mg/m2 D1 doxorubicin 50 mg/m2 D1 vincristine 1.4 mg/m2 D1 prednisone 100 mg D1-D5
  2. Phase II Bortezomib 1.6 mg/m2 CHOP,every 2 weeks cyclophosphamide 750 mg/m2 D1 doxorubicin 50 mg/m2 D1 vincristine 1.4 mg/m2 D1 prednisone 100 mg D1-D5
Period: Overall Study
Arm/Group | Bortezomib + CHOP Every 2 Weeks
Started | 49 (Phase I (9) + Phase II (40))
Completed | 49 (Phase I (9) + Phase II (40))
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bortezomib + CHOP Every 2 Weeks: CHOP; cyclophosphamide, doxorubicin, vincristine, and prednisone
Arm/Group | Bortezomib + CHOP Every 2 Weeks
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 24
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieved Complete Response
Description: All patients,9 patients of phase I study and 40 patietns in phase II stuay, were assessed with International Working Group response criteria assessed by CT; Complete Response (CR), Disappearance of all detectable clinical and radiographic evidence of disease and diappearance of all disease-related symptoms.
Time Frame: 14 weeks
Measure: Number; unit: participants
Arm/Group | Bortezomib + CHOP Every 2 Weeks
Number analyzed (Participants) | 49
participants | 32 [65.2 to 89.5]

2. Secondary Outcome: Number of Patients Who Experienced Adverse Events
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Bortezomib + CHOP Every 2 Weeks
Number analyzed (Participants) | 49
participants | 49

ADVERSE EVENTS:
Arm/Group | Bortezomib + CHOP Every 2 Weeks
Serious Adverse Events (participants affected / at risk) | 22/49
Other Adverse Events (participants affected / at risk) | 27/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Bortezomib + CHOP Every 2 Weeks (N=49)
abdominal pain (Gastrointestinal disorders) | 4/40 (4)
constipation (Gastrointestinal disorders) | 0/40 (0)
diarrhea (Gastrointestinal disorders) | 4/40 (4)
fatigue (Metabolism and nutrition disorders) | 2/40 (2)
hyperglycemia (Endocrine disorders) | 4/40 (4)
vomiting (Gastrointestinal disorders) | 4/40 (4)
sensory neuropathy (Nervous system disorders) | 11/40 (11)
motor neuropathy (Nervous system disorders) | 3/40 (3)
anemia (Blood and lymphatic system disorders) | 22/40 (22)
neutropenia (Blood and lymphatic system disorders) | 14/40 (14)
feberile neutropenia (Blood and lymphatic system disorders) | 7/40 (15)
thrombocytopenia (Blood and lymphatic system disorders) | 13/40 (13)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Bortezomib + CHOP Every 2 Weeks (N=49)
abdominal pain (Gastrointestinal disorders) | 27/40 (27)
anorexia (Gastrointestinal disorders) | 25/40 (26)
constipation (Gastrointestinal disorders) | 23/40 (24)
diarrhea (Gastrointestinal disorders) | 21/40 (22)
fatigue (Metabolism and nutrition disorders) | 23/40 (25)
nausea (Gastrointestinal disorders) | 12/40 (21)
nausea (Gastrointestinal disorders) | 11/40 (20)
vomiting (Gastrointestinal disorders) | 16/40 (20)
sensory neuropathy (Nervous system disorders) | 22/40 (27)
motor neuropathy (Nervous system disorders) | 17/40 (21)
anemia (Blood and lymphatic system disorders) | 11/40 (19)
neutropenia (Blood and lymphatic system disorders) | 12/40 (15)
febrile neutropenia (Infections and infestations) | 6/40 (7)
thrombocytopenia (Blood and lymphatic system disorders) | 15/40 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No